CLINICAL TRIAL: NCT01104480
Title: Efficacy of Tocilizumab in a Patient With Relapsing Polychondritis
Brief Title: Tocilizumab for Relapsing Polychondritis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Tocilizumab was licenced in Canada for children, so the study was not necessary
Sponsor: McMaster Children's Hospital (Other)
Responsible Party: Principal Investigator, Dr Maggie Larche, Associate professor, McMaster Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP2010
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Relapsing Polychondritis
Keywords: Relapsing Polychondritis; Unremitting; Inflammation; IL6
MeSH Terms: conditions — Polychondritis, Relapsing; Inflammation | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab 8mg/kg every 2 weeks given by IV infusion
  Other Names: Actemra

SUMMARY:
This is a study for one patient with severe relapsing polychondritis which has been unresponsive to other more conventional medications including prednisone, methotrexate, anakinra and TNF inhibitors. Tolerability, and efficacy of the drug, Tocilizumab will be monitored by clinical assessment and bloodwork.

ELIGIBILITY:
Inclusion Criteria:

* A single patient with unremitting inflammatory relapsing polychondritis

Exclusion Criteria:

* As this is a study in a single patient, there are no exclusions

Ages: 12 Years to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Tocilizumab | 2 years
  Inhibition of inflammatory markers Improvement in symptoms and signs

SECONDARY OUTCOMES:
Safety of Tocilizumab | 2 years
  Monitoring of serum lipids and liver function tests

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Larché, MD, PhD, Principal Investigator — McMaster University and Children's Hospital
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada